CLINICAL TRIAL: NCT00597805
Title: A Prospective Study of Quality of Life in Patients Undergoing Pelvic Exenteration
Brief Title: Quality of Life in Patients Undergoing Total Pelvic Exenteration
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 05-001
Record Dates: First submitted 2008-01-09; First posted 2008-01-18 (Estimated); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Total Exenteration; Anterior or Posterior Pelvic Exenteration; Gynecologic Malignancies; Colorectal Malignancies; Urologic Malignancies
MeSH Terms: interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients scheduled for a total, anterior or posterior pelvic exenteration
  Interventions: Behavioral: questionnaires/interviews

INTERVENTIONS:
Behavioral: questionnaires/interviews — All patients who agree to participate will be interviewed for a baseline quality of life assessment prior to surgery. A brief in hospital interview will follow in the peri-operative period. In the ensuing months, patients will be interviewed at approximately 3, 6 and 12 months post-operatively (eg: 3 month interview will be done between 8-16 weeks and 6 month interview between 20-28 months post-operatively). Annual interviews in years two through five will be employed to determine areas for future study and solicit narrative on transition toward cancer survivorship.

SUMMARY:
The purpose of this study is to learn more about the personal experiences of patients who are treated with pelvic exenteration surgery. Pelvic exenteration is a surgical procedure in which the pelvic organs including the reproductive organs, bladder and/or rectum are removed. We would like to understand more about the physical, emotional, educational, and sexual needs of patients who are treated with this surgery. We will use what we learn from this study to help find better ways of preparing patients for this type of surgery. This will also allow us to be more helpful to patients' needs after surgery.

DETAILED DESCRIPTION:
This protocol represents the first study to comprehensively evaluate QOL in a mixed population of male and female patients treated with total, anterior or posterior pelvic exenteration. This unique approach to QOL assessment which is both domain-centered and able to emphasize individual differences through the C-SHIP model has the potential to set the standard for evaluating QOL in patients who undergo extensive pelvic surgery. The longitudinal design of this study facilitates the documentation of patients'responsiveness to change. By analyzing participants' responses at intervals we will be able to document the redefinition of life goals which occurs as patients adapt to their new health status. The data and analysis completed in first three years of this study will be used to generate further hypotheses for future investigation.

ELIGIBILITY:
Inclusion Criteria:

* All patients (male and female) who are scheduled to undergo total, anterior or posterior pelvic exenteration for pelvic malignancies arising in gynecologic, colorectal or urologic organs are eligible for participation in the study. Anterior or posterior pelvic exenteration must involve formation of a permanent ostomy (urostomy or colostomy).
* Participants must be able to speak and read English proficiently.
* Participants must be able to provide written informed consent.
* Patients must be 18 years of age or older to enroll.

Exclusion Criteria:

* Subjects may be excluded or withdrawn from the study based on the following criteria.
* Development of a cognitive or psychiatric deficit resulting in an inability to provide meaningful informed consent
* Inability to speak or read in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MSKCC's Clinics and Moffitt Cancer Center, Tampa, Florida
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2005-01 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2024-12-12 (Actual)

PRIMARY OUTCOMES:
To characterize the extent of physical and psychological stress, and overall quality of life in patients undergoing total, anterior or posterior pelvic exenteration. | conclusion of study

SECONDARY OUTCOMES:
To determine how patients ratings of the specific QOL domains predict response to surgery, (ie; QOL, level of stress, function and symptoms). | conclusion of study

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Chi, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org